CLINICAL TRIAL: NCT00851344
Title: A Randomised, Double-blind, Placebo-controlled, 4-period Incomplete Block Crossover Study of Single Oral Dose GSK835726 (100mg, 50mg, 10mg), Cetirizine (10mg) and Placebo to Evaluate the Efficacy and Safety Using an Environmental Challenge Chamber in Male Subjects With Seasonal Allergic Rhinitis
Brief Title: Allergen Challenge Chamber Study With Single Dose Oral GSK835726 Compared With Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 110163
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Proof-of-Concept; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — GSK 835726; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- GSK835726 (10mg) (Active Comparator): 10mg oral dose
  Interventions: Drug: GSK835726 (10mg)
- GSK835726 (50mg) (Active Comparator): 50mg oral dose
  Interventions: Drug: GSK835726 (50mg)
- GSK835726 (100mg) (Active Comparator): 50mg oral dose
  Interventions: Drug: GSK835726 (100mg)
- Cetirizine 10mg (Active Comparator): 10mg cetirizine as active comparator
  Interventions: Drug: Cetirizine (10mg)
- placebo (Placebo Comparator): placebo tablet
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSK835726 (10mg) — GSK835726 (10mg) tablet
  Arms: GSK835726 (10mg)
Drug: GSK835726 (50mg) — GSK835726 (50mg) tablet
  Arms: GSK835726 (50mg)
Drug: GSK835726 (100mg) — GSK835726 (100mg) tablet
  Arms: GSK835726 (100mg)
Drug: Cetirizine (10mg) — Cetirizine (10mg) tablet as positive control
  Arms: Cetirizine 10mg
Other: Placebo — Placebo to match active
  Arms: placebo

SUMMARY:
A randomised, double-blind, placebo-controlled, 4-period incomplete block crossover study of single oral dose GSK835726 (100mg, 50mg, 10mg), Cetirizine (10mg) and placebo to evaluate the efficacy and safety using an Environmental challenge chamber in male subjects with seasonal allergic rhinitis

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy apart from seasonal allergic rhinitis, as determined by a physician. Can have mild asthma.
* Male
* Aged 18 - 60
* Weight 50kg+, BMI 19-32 kg/m2
* Exhibit response to Challenge Chamber and skin prick test.
* Non-smoker
* Capable of giving informed consent

Exclusion Criteria:

* No nasal structural abnornmality/polyposis, surgery, infection.
* any respiratory disease, other than mild asthma or seasonal allergic rhinitis
* participated in another clinical study within 30 days.
* Subject has donated a unit of blood within 1 month
* Use of prescription or non-prescription drugs, including vitamins and st john's wort within 7 days of trial.
* History of sensitivty to drug
* History of alcohol/drug abuse within 12 months.
* Positive Hepatitis B antibody test
* Positive HIV antibody test
* Risk of non-compliance with study protocol
* Perenial allergic rhinitis
* Administration of oral, injectable or dermal corticosteriods within 8 weeks, intranasal or inhaled within 3 weeks.
* Past or present disease that may affect outcome, as judge by investigator
* Specific Immunotherapy within 2 years

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total nasal symptom score 0-4 hours post dose | 0-4 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Daley-Yates P, Ambery C, Sweeney L, Watson J, Oliver A, McQuade B. The efficacy and tolerability of two novel H(1)/H(3) receptor antagonists in seasonal allergic rhinitis. Int Arch Allergy Immunol. 2012;158(1):84-98. doi: 10.1159/000329738. Epub 2011 Dec 29. PMID 22212854
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 110163 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110163 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110163 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110163 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110163 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110163 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110163 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register